CLINICAL TRIAL: NCT01044446
Title: Effect of Icodextrin on the Treatment Outcome of Peritoneal Dialysis Patients
Brief Title: Effect of Icodextrin on the Treatment Outcome of Peritoneal Dialysis Patients During Acute Peritonitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chow Kai Ming, Associate Consultant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2009.481
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Peritonitis
Keywords: peritoneal dialysis; peritonitis; CAPD; end-stage renal disease; peritonitis outcome and ultrafiltration
MeSH Terms: conditions — Peritonitis; Kidney Failure, Chronic | interventions — Icodextrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Icodextrin (Experimental): peritoneal dialysate
  Interventions: Drug: Icodextrin
- Glucose-based dialysate (Active Comparator): peritoneal dialysate
  Interventions: Drug: glucose-based peritoneal dialysate

INTERVENTIONS:
Drug: Icodextrin — one exchange daily
  Arms: Icodextrin
Drug: glucose-based peritoneal dialysate — original exchange frequency
  Arms: Glucose-based dialysate

SUMMARY:
The objective of the present study is to evaluate the a prior hypothesis that treatment with icodextrin during acute peritonitis would improve the treatment outcomes of peritonitis complicating peritoneal dialysis. The safety and effectiveness of icodextrin for decreasing glucose exposure, extent and severity of peritonitis will be evaluated in the setting of acute peritonitis complicating peritoneal dialysis among patients who are not receiving icodextrin.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or older on peritoneal dialysis, who develop clinical evidence of peritonitis
* stable peritoneal dialysis with Baxter connection system
* willingness to give written consent and comply with the study protocol

Exclusion Criteria:

* already on icodextrin dialysate prior to acute presentation with peritonitis
* known allergy or hypersensitivity to icodextrin, starch or have a glycogen storage disease
* participation in another interventional study within last 30 days of randomization
* history of a psychological illness or condition that would interfere with the patient's ability to understand the requirement of the study and/or comply with the study procedures

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-01; Primary Completion 2012-08 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
peritoneal dialysate total white cell count on day 3 of acute peritonitis | day 3

SECONDARY OUTCOMES:
need of additional hypertonic exchanges, ultrafiltration volumes according to patient diary, fluid control as denoted by changes in body weight, and the timing of peritonitis resolution | within the period of peritonitis treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Chinese University of Hong Kong, Shatin, New Territories, Hong Kong

REFERENCES:
- [Derived] Chow KM, Szeto CC, Kwan BC, Pang WF, Ma T, Leung CB, Law MC, Li PK. Randomized controlled study of icodextrin on the treatment of peritoneal dialysis patients during acute peritonitis. Nephrol Dial Transplant. 2014 Jul;29(7):1438-43. doi: 10.1093/ndt/gfu033. Epub 2014 Feb 26. PMID 24578470